CLINICAL TRIAL: NCT05093556
Title: Interactive CBT for Headache And Relaxation Training (iCHART)
Brief Title: Interactive CBT for Headache And Relaxation Training
Acronym: iCHART
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in vendor security protocols would have necessitated changing platforms and rebuilding entire IVR platform which would have delayed patient recruitment and introduced heterogeneity across subjects using current and new platforms
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG001
Record Dates: First submitted 2021-09-22; First posted 2021-10-26 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Post-Traumatic Headache
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iCHART - Interactive CBT for Headache And Relaxation Training (Experimental): 10 week interactive-voice response technology (IVR) based cognitive behavioral therapy for headache
  Interventions: Behavioral: iCHART - Interactive CBT for Headache And Relaxation Training

INTERVENTIONS:
Behavioral: iCHART - Interactive CBT for Headache And Relaxation Training — IVR based cognitive behavioral therapy for headache

SUMMARY:
This mixed-methods pilot study aims to evaluate the feasibility, acceptability, and preliminary effectiveness of iCHART (Interactive CBT for Headache And Relaxation Training), an interactive voice response (IVR) based delivery of cognitive behavioral therapy for Veterans with post-traumatic headache. Participants will receive iCHART treatment through the IVR system over a period of 10 weeks, which will include an automated daily assessment of patient-reported outcomes, retrieval of fortnightly tailored feedback from a study therapist, and additional weekly one-way motivational enhancement messaging. Delivery of traditional evidence-based behavioral treatments for headache management through technology-based interventions, such as IVR may ultimately increase much needed access to these treatments and allow patients to receive care at a time that is convenient for them.

DETAILED DESCRIPTION:
Headache disorders are prevalent and highly disabling chronic neurological pain conditions, especially among women and people with traumatic brain injury, yet remain underdiagnosed and undertreated. Cognitive behavioral therapy for headache is an evidence-based psychological treatment that is effective in reducing headache frequency and severity, addressing psychiatric comorbidities, and improving an individual's quality of life, yet it remains hugely underutilized and inaccessible to many. Delivery of traditional evidence-based behavioral treatments for headache management through technology-based interventions may ultimately increase much needed access to these treatments. Interactive voice response (IVR) is an automated telephone-based technology where people receive tailored messaging which allows them to track symptoms, target behavior change, and engage in disease self-management. This mixed-methods pilot study aims to evaluate the feasibility, acceptability, and preliminary effectiveness of iCHART (Interactive CBT for Headache And Relaxation Training), an IVR-based delivery of cognitive behavioral therapy for Veterans with headache.

Participants will be thirty-five Veterans receiving care within VA Connecticut Healthcare System, who are diagnosed with post-traumatic headache. All eligible participants will complete an initial intake interview and a 28-day electronic headache diary. Following the baseline assessment period, eligible participants will then receive iCHART treatment through the IVR system over a period of 10 weeks, which will include an automated daily assessment of patient-reported outcomes, retrieval of fortnightly tailored feedback from a study therapist, and additional weekly one-way motivational enhancement messaging. Participants will access a patient workbook via the iCHART study website and iCHART providers will visualize patient-reported data through the secure iCHART provider dashboard. Assessment measures will be completed at baseline, immediately post-treatment completion, and one month post-treatment completion. Analysis of primary and secondary outcome measures will employ mixed methods.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of post-traumatic headache disorder (migraine and/or tension-type subtype)
* Frequency of ≥4 headache days per month
* Primary pain complaint of headache
* Access to a touchtone telephone and computer/tablet

Exclusion Criteria:

* Non-English speaking
* Non-Veteran
* Receiving hospice or palliative care
* Sensory deficits that would impair participation in the IVR telephone calls
* Significant cognitive impairment
* Inpatient psychiatric hospitalization for any psychiatric or substance use diagnosis in the past 30 days from screening
* Active psychotic symptoms, suicidality, or severe depressive symptoms
* Suicidal and/or homicidal ideation in the past 6 months from screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change in headache days | Baseline and week 14
  Daily self-reported headache days

SECONDARY OUTCOMES:
Change in headache-related disability | Baseline and week 14
  Headache Disability Inventory (HDI) is a 25-item self-report questionnaire that assesses both emotional and functional impact of headache on daily activities. Item response options include "yes", "sometimes", and "no." Total scores range from 0 to 100. Higher scores indicate higher levels of reported disability.
Change in headache-related disability | Baseline and week 14
  Migraine Disability Assessment (MIDAS) is a 5-item, self-report measure of life disruption due to headache. Cut points represent thresholds for little or no disability (0-5), mild disability (6-10), moderate disability (11-20), and severe disability (21+).

OTHER OUTCOMES:
Veterans RAND 12-item Health Survey (VR-12) | Baseline, week 10, and week 14
  A 12-item, self-report measure of health-related quality life in terms of physical and mental health domains. Scores are summed into a physical health and mental health summary score and standardized using a T-score metric with a mean of 50 and a standard deviation of 10.
Patient Health Questionnaire 8-item (PHQ-8) | Baseline, week 10, and week 14
  An 8-item, self-report measure of depressive symptom severity based on DSM criteria. Items are rated from 0 to 3 (0 = not at all to 3 = nearly every day). Total scores range from 0 to 27. Cut points represent thresholds for non-minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19), and severe (20-27) depression.
Generalized Anxiety Disorder Screener (GAD-7) | Baseline, week 10, and week 14
  A 7-item, self-report measure of anxiety. Items are rated from 0 to 3 (0 = not at all to 3 = nearly every day). Total scores range from 0 to 21. Cut points represent thresholds for none-minimal (0-4), mild (5-9), moderate (10-14) and severe (15-21).
Post-Traumatic Stress Disorder Checklist (PCL) | Baseline, week 10, and week 14
  A 17-tem, self-report measure of symptoms of PTSD based on Diagnostic and Statistical Manual (DSM) criteria. Items are rated from 0 to 4 (0= Not at all to 4 = Extremely). Total scores range from 17-85.
Insomnia Severity Index (ISI) | Baseline, week 10, and week 14
  A 5-item self-report measure of symptoms of insomnia. Total scores range from 0 to 28. Cut points represent thresholds for no clinically significant insomnia (0-7), subthreshold insomnia (8-14), clinical insomnia (moderately severe) (15-21), clinical insomnia (severe) (22-28).
Headache Pain Catastrophizing Scale (HPCS) | Baseline, week 10, and week 14
  A modified version of the Pain Catastrophizing Scale (use of word headache vs. pain in the questions). The HPCS is a 13-item self-report measure of catastrophic thinking related to headache. Items are rated from 0 to 4 (0= not at all to 4 - all the time). Total scores range from 0 to 52, with subscale scores for rumination, magnification, and helplessness.
Headache Management Self-Efficacy Scale (HMSE) | Baseline, week 10, and week 14
  A 25-item self-report questionnaire related to a person's confidence in their ability to manage their headache symptoms. Items range from 1 to 7 (1=strongly disagree to 7 = strongly disagree). Total scores range from 25 to 175
Patient Global Perception of Change (PGPC) | Week 10
  single item scale measures the participant's perception of improvement since the start of the study. Participants respond to the single item on a 7-point scale (1 = very much improved to 7 = very much worse). This measure shows good psychometric properties.
Client Satisfaction Questionnaire-8 (CSQ-8) | Week 10
  An 8-item self-report measure of treatment acceptability and satisfaction with mental health treatment. Items are coded on a 4-point scale. Total scores are calculated by summing up items, with scores ranging from 8 to 32
System Usability Scale (SUS) | Week 10
  A 10-item measure of treatment acceptability. The SUS assesses participant perceived usability of technology systems. Response options range from 1 to 5, with 50% of the items being positively worded and 50% negatively worded. Scores are converted to an overall score from 0 to 100. Higher scores indicate higher perceived usability
Acceptability of Intervention (AIM) | Week 10
  A 4-item measure of treatment acceptability. Items are score on a 5-point scale. Scores are a calculated mean. Higher scores indicate greater acceptability
Structured Assessment of Feasibility Questionnaire (SAFE) | Week 10
  A 16-item measure of feasibility of mental health services, organized into two sections. The first eight questions assess barriers to implementation, the final eight assess facilitators to implementation. Items are rated as either yes, partial, no, or unable to rate, with each individual item attended to. It is recommended against using a summary score, since items within the sale may have unequal weight.
Feasibility of Intervention Measure (FIM) | Week 10
  A 4-item measure of feasibility. Items are rated on a 5-point Likert scale. Scores are a calculated mean. Higher scores indicate greater feasibility

CONTACTS AND LOCATIONS:
Overall Officials: Amy Grinberg, PhD, Principal Investigator — VA Connecticut Healthcare System
Locations (1):
- VACHS, West Haven, Connecticut, United States

REFERENCES:
- [Derived] Grinberg AS, Rogers DG, Datre O, Anthony S, Clark SW, Takagishi SC, Seng E, Fenton BT, Ney JP, Sico JJ. Interactive CBT for headache and relaxation training (iCHART): Single-arm pilot trial of cognitive behavioral therapy for veterans with post-traumatic headache. Cephalalgia. 2025 Jul;45(7):3331024251351598. doi: 10.1177/03331024251351598. Epub 2025 Jul 14. PMID 40657938